CLINICAL TRIAL: NCT01432730
Title: A Study to Assess the Efficacy of AF-219, a P2X3 Receptor Antagonist, in Subjects With Chronic Cough (EPiCC)
Brief Title: A Study to Assess the Efficacy of Gefapixant (MK-7264/AF-219), in Participants With Chronic Cough (MK-7264-006)
Acronym: EPICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-006; AF219-006 (Other: Afferent Pharmaceuticals); MK-7264-006 (Other: Merck); 2010-024283-18 (EudraCT Number)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gefapixant 600 mg>Placebo (Experimental): Gefapixant, 600 mg, twice daily (BID), taken orally for 2 weeks followed by a 2-week washout period and then placebo to gefapixant, BID, taken orally for 2 weeks.
  Interventions: Drug: Gefapixant; Drug: Placebo
- Placebo>Gefapixant 600 mg (Experimental): Placebo to gefapixant BID, taken orally for 2 weeks followed by a 2-week washout period and then gefapixant, 600 mg, BID, taken orally for 2 weeks.
  Interventions: Drug: Gefapixant; Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant — Oral tablets, BID
  Other Names: AF-219; MK-7264
Drug: Placebo — Oral tablets, BID

SUMMARY:
This is a randomised, double-blind, placebo-controlled, crossover, single centre study of gefapixant (AF-219/MK-7264) in participants with idiopathic or treatment resistant chronic cough designed to evaluate the effectiveness of gefapixant in reducing daytime objective cough frequency.

ELIGIBILITY:
Inclusion Criteria:

* History of cough for more than 8 weeks
* Normal chest radiograph
* Idiopathic or treatment resistant cough (idiopathic defined as a cough for which no objective evidence of an underlying trigger can be determined after investigation or a cough that is unresponsive to 8 weeks of targeted treatment for identified underlying triggers including reflux disease, asthma and post-nasal drip [treatment-resistant]).

Exclusion Criteria:

* Current smoker
* Individuals who have given up smoking within the past 6 months, or those with >20 pack-year smoking history
* Treatment with an angiotensin-converting-enzyme inhibitor (ACE-inhibitor) as the potential cause of a participant's cough, or requiring treatment with an ACE-inhibitor during the study or within 4 weeks prior to Day 0
* Forced Expiratory Volume (FEV1)/Forced Vital Capacity (FVC) <60%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09-22 (Actual); Primary Completion 2013-02-07 (Actual); Study Completion 2013-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Abdulqawi R, Dockry R, Holt K, Layton G, McCarthy BG, Ford AP, Smith JA. P2X3 receptor antagonist (AF-219) in refractory chronic cough: a randomised, double-blind, placebo-controlled phase 2 study. Lancet. 2015 Mar 28;385(9974):1198-205. doi: 10.1016/S0140-6736(14)61255-1. Epub 2014 Nov 25. PMID 25467586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 participants were enrolled and randomized from a single center.
Groups:
- Gefapixant 600 mg>Placebo: Gefapixant, 600 mg, twice daily (BID), taken orally for 2 weeks in Period 1 followed by a 2-week washout period and then placebo, BID, taken orally for 2 weeks in Period 2
- Placebo>Gefapixant 600mg: Placebo BID, taken orally for 2 weeks in Period 1 followed by a 2-week washout period and then gefapixant, 600 mg, BID, taken orally for 2 weeks in Period 2
Period: Period 1
Arm/Group | Gefapixant 600 mg>Placebo | Placebo>Gefapixant 600mg
Started | 12 | 12
Completed | 10 | 12
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Period 2
Arm/Group | Gefapixant 600 mg>Placebo | Placebo>Gefapixant 600mg
Started | 10 | 12
Completed | 10 | 8
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- All Participants: Gefapixant, 600 mg, BID, taken orally for 2 weeks in Period 1 followed by a 2-week washout period and then placebo to gefapixant, BID, taken orally for 2 weeks in Period 2 OR Placebo to gefapixant, BID, taken orally for 2 weeks in Period 1 followed by a 2-week washout period and then gefapixant, 600 mg, BID, taken orally for 2 weeks in Period 2
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daytime Objective Cough Frequency
Description: Daytime Objective Cough Frequency (per hour) is the total number of cough events during the monitoring period (in general, 24-hr interval) the participant is awake divided by the total duration (in hours) for the monitoring period the participants is awake. 24-hour sound recordings were collected using a digital recording device. Change from baseline in awake cough frequency = (post-treatment awake cough frequency - baseline awake cough frequency). A negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency.
Time Frame: Baseline (Day 0) and Day 14 of each study period
Population: Analysis population consisted of all participants for Periods 1 and 2 who were randomized, received at least 1 dose of study drug, were compliant with the study procedure and had available data for this outcome measure.
Measure: Log Mean (Standard Error); unit: Coughs/hour
Groups:
- Gefapixant 600 mg: Gefapixant 600 mg twice daily (BID) taken orally for 2 weeks
- Placebo: Placebo BID taken orally for 2 weeks
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 19 | 21
Coughs/hour | -0.5365 (0.1718) | 0.0523 (0.0462)
Statistical Analysis 1: Comparison: Gefapixant 600 mg vs Placebo; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mixed model included terms for treatment sequence, participant within sequence, treatment & period. Average & period baseline covariates included; Log mean difference (Active - Placebo) = -0.6027, 95% CI 2-sided [-0.9049 to -0.3005]

2. Secondary Outcome: Change From Baseline of Daytime Cough Severity Score Using a Visual Analogue Scale (VAS)
Description: Cough Severity VAS: scored from 0 to 100 using a 10 mm visual analogue scale with 0 at 0mm and 100 at 100mm with 0 representing no cough and 100 the most severe cough. Change from baseline in daytime cough severity = (post-treatment daytime cough severity - baseline daytime cough severity). A negative result indicates a decrease in cough severity, while a positive result indicates an increase in cough severity.
Time Frame: Baseline (Day 0) and Day 15 of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 20 | 21
Score on a scale | -21.5 (35.65) | -0.7 (19.01)
Statistical Analysis 1: Comparison: Gefapixant 600 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mixed effect model fitting terms for treatment sequence, participant within sequence, treatment, and period; Mean Difference (Final Values) = -25.57, 95% CI 2-sided [-41.53 to -9.62]

3. Secondary Outcome: Change From Baseline in Nighttime Objective Cough Frequency
Description: Nighttime Objective Cough Frequency = Total number of cough events during the monitoring period the participant is asleep divided by the total duration (in hours) for the monitoring period the participant is asleep. 24 hour sound recording were collected with a digital recording device. Change from baseline in nighttime cough frequency = (post-treatment nighttime cough frequency - baseline nighttime cough frequency). A negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency.
Time Frame: Baseline (Day 0) and Day 14 of each study period
Population: as for outcome 1
Measure: Log Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 18 | 20
Coughs/hour | -0.3452 (0.2314) | 0.0690 (0.1767)
Statistical Analysis 1: Comparison: Gefapixant 600 mg vs Placebo; Test type: Superiority; p = 0.057, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Log mean difference (Active - Placebo) = -0.4212, 95% CI 2-sided [-0.8568 to 0.01438]

4. Secondary Outcome: Change From Baseline of Nighttime Cough Severity Score Using a Visual Analogue Scale (VAS)
Description: Cough Severity VAS: scored from 0 to 100 using a 10 mm visual analogue scale with 0 at 0mm and 100 at 100mm with 0 representing no cough and 100 the most severe cough. Change from baseline in nighttime cough severity = (post-treatment nighttime cough severity - baseline nighttime cough severity). A negative result indicates a decrease in cough severity, while a positive result indicates an increase in cough severity.
Time Frame: Baseline (Day 0) and Day 15 of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 20 | 21
Score on a scale | -16.1 (27.71) | -3.7 (22.05)
Statistical Analysis 1: Comparison: Gefapixant 600 mg vs Placebo; Test type: Superiority; p = 0.172, Mixed Models Analysis; Mixed effect model fitting terms for treatment sequence, participant within sequence, treatment, and period; Mean Difference (Final Values) = -8.53, 95% CI 2-sided [-20.93 to 3.87]

5. Secondary Outcome: Change From Baseline of 24-hour Objective Cough Frequency
Description: Total (0-24 hours) Objective Cough Frequency = Total number of cough events during the monitoring period divided by the total duration (in hours, i.e., 24 hours mostly) for the monitoring period. 24-hour sound recordings were collected using a digital recording device. A negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency.
Time Frame: 24 hours at Baseline (Day 0) and Day 14 of each study period
Population: as for outcome 1
Measure: Log Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 18 | 20
Coughs/hour | -0.5562 (0.1795) | 0.0298 (0.0459)
Statistical Analysis 1: Comparison: Gefapixant 600 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Log mean difference (Active - Placebo) = -0.582, 95% CI 2-sided [-0.8934 to -0.2707]

6. Secondary Outcome: Global Rating of Change Score for Cough Frequency
Description: At the end of each study period, participants were asked to complete the global rating of change scale questionnaire. The participants were asked to record whether their cough frequency was "worse", "about the same", or "better". If better or worse, the participants were then asked "by how much" with a 7-category rating scale. Therefore, a 15-point ordered scale was used (1=minimum, a very great deal better to 15=maximum, a very great deal worse with a score of 8=indicating no change).
Time Frame: Day 15 of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 24 | 22
Score on a scale | 5.83 (4.96) | 8.32 (2.28)
Statistical Analysis 1: Comparison: Gefapixant 600 mg vs Placebo; Test type: Superiority; p = 0.033, Mixed Models Analysis; Mixed effect model fitting terms for treatment sequence, participant within sequence, treatment, and period; Mean Difference (Final Values) = -2.538, 95% CI 2-sided [-4.849 to -0.227]

7. Secondary Outcome: Global Rating of Change Score for Cough Severity
Description: At the end of each study period, participants were asked to complete the global rating of change scale questionnaire. The participants were asked to record whether their cough severity was "worse", "about the same", or "better". If better or worse, the participants were then asked "by how much" with a 7-category rating scale. Therefore, a 15-point ordered scale was used (1=minimum, a very great deal better to 15=maximum, a very great deal worse with a score of 8=indicating no change).
Time Frame: Day 15 of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 24 | 22
Score on a scale | 6.00 (4.94) | 8.23 (2.25)
Statistical Analysis 1: Comparison: Gefapixant 600 mg vs Placebo; Test type: Superiority; p = 0.049, Mixed Models Analysis; Mixed effect model fitting terms for treatment sequence, participant within sequence, treatment, and period; Median Difference (Final Values) = -2.267, 95% CI 2-sided [-4.523 to -0.010]

8. Secondary Outcome: Change From Baseline in Cough-specific Quality of Life Questionnaire (CQLQ)
Description: The CQLQ Questionnaire included 28 items that described negative aspects of quality of life specific to chronic cough. Subscales include: Physical complaints, Psychosocial issues, Functional abilities, Emotional wellbeing, Extreme physical complaints, and Personal safety fears. Participants indicated their degree of agreement with each statement on a 4 point scale (1 = strongly disagree; 2 = disagree; 3 = agree; 4 = strongly agree). CQLQ scores (28 for least impact, 112 for highest impact) used a mixed effect model with terms for treatment sequence, participant within sequence, treatment, and period. Change from baseline in CQLQ scores = (posttreatment CQLQ scores - baseline CQLQ scores). A negative result indicates a decrease in CQLQ scores (lowest cough impact on health-related quality of life), while a positive result indicates an increase in CQLQ scores (highest cough impact on health-related quality of life).
Time Frame: Baseline (Day 0) and Day 15 of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 19 | 17
Score on a scale | -10.8 (14.23) | -1.4 (6.48)
Statistical Analysis 1: Comparison: Gefapixant 600 mg; Test type: Superiority; p = 0.018, Mixed Models Analysis; Mixed effect model fitting terms for treatment sequence, participant within sequence, treatment, and period; Mean Difference (Final Values) = -9.237, 95% CI 2-sided [-16.759 to -1.716]

9. Secondary Outcome: Change From Baseline in Urge to Cough Questionnaire (UtCQ) 100 mm Visual Analogue Scale
Description: UtCQ is determined through the use of a 100mm visual analogue scale (VAS) (ranging between 0 for "no urge to cough" and 100 for "severe urge to cough"). Change from baseline in UtCQ scores = (post-treatment UtCQ scores - baseline UtCQ scores). A negative result indicates a decrease in UtCQ scores (lowest impact), while a positive result indicates an increase in UtCQ scores (highest impact).
Time Frame: Baseline (Day 0) and Day 15 of each study period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 24 | 20
Score on a scale | -27.2 (42.07) | -6.5 (28.59)
Statistical Analysis 1: Comparison: Gefapixant 600 mg vs Placebo; Test type: Superiority; p = 0.035, Mixed Models Analysis; Mixed effect model fitting terms for treatment sequence, participant within sequence, treatment, and period; Mean Difference (Final Values) = -21.25, 95% CI 2-sided [-40.96 to -1.54]

10. Other Pre Specified Outcome: Baseline Daytime Cough Frequency
Description: Daytime Objective Cough Frequency (per hour) is the total number of cough events during the monitoring period (in general, 24-hr interval) the participant is awake divided by the total duration (in hours) for the monitoring period the participants is awake. 24-hour sound recordings were collected using a digital recording device.
Time Frame: Baseline (Day 0) of each study period
Population: Analysis population consisted of all participants for Periods 1 and 2 who were randomized, were compliant with the study procedure and had available data at baseline for daytime cough frequency.
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 19 | 21
Coughs/hour | 37.09 (32.23) | 65.45 (163.36)

11. Other Pre Specified Outcome: Baseline Daytime Cough Severity Score Using a Visual Analogue Scale (VAS)
Description: Cough Severity VAS is scored from 0 to 100 using a 10 mm visual analogue scale with 0 at 0mm and 100 at 100mm with 0 representing no cough and 100 the most severe cough.
Time Frame: Baseline (Day 0) of each study period
Population: Analysis population consisted of all participants for Periods 1 and 2 who were randomized, were compliant with the study procedure and had available data at baseline for daytime cough severity.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 20 | 21
Score on a scale | 48.8 (20.73) | 52.7 (16.10)

12. Other Pre Specified Outcome: Baseline Nighttime Objective Cough Frequency
Description: Nighttime Objective Cough Frequency is the total number of cough events during the monitoring period the participant is asleep divided by the total duration (in hours) for the monitoring period the participant is asleep. 24 hour sound recording were collected with a digital recording device.
Time Frame: Baseline (Day 0) of each study period
Population: Analysis population consisted of all participants for Periods 1 and 2 who were randomized, were compliant with the study procedure and had available data at baseline for nighttime cough frequency.
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 18 | 20
Coughs/hour | 4.34 (7.79) | 7.78 (23.80)

13. Other Pre Specified Outcome: Baseline Nighttime Cough Severity Score Using a Visual Analogue Scale (VAS)
Description: Nighttime cough severity was scored from 0 to 100 using a 10 mm visual analogue scale with 0 at 0mm and 100 at 100mm with 0 representing no cough and 100 the most severe cough.
Time Frame: Baseline (Day 0) of each study period
Population: Analysis population consisted of all participants for Periods 1 and 2 who were randomized, were compliant with the study procedure and had available data at baseline for nighttime cough severity.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 20 | 21
Score on a scale | 31.5 (23.86) | 28.8 (24.88)

14. Other Pre Specified Outcome: Baseline 24-Hour Objective Cough Frequency
Description: Total (0-24 hours) Objective Cough Frequency = Total number of cough events during the monitoring period divided by the total duration (in hours, i.e., 24 hours mostly) for the monitoring period. 24-hour sound recordings were collected using a digital recording device.
Time Frame: Baseline (Day 0) of each study period
Population: Analysis population consisted of all participants for Periods 1 and 2 who were randomized, were compliant with the study procedure and had available data at baseline for 24-hour objective cough frequency.
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 18 | 20
Coughs/hour | 26.63 (22.63) | 44.70 (105.16)

15. Other Pre Specified Outcome: Baseline Cough-specific Quality of Life Questionnaire (CQLQ)
Description: as for outcome 8
Time Frame: Baseline (Day 0) of each study period
Population: Analysis population consisted of all participants for Periods 1 and 2 who were randomized, were compliant with the study procedure and had available data at baseline for CQLQ.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 19 | 17
Score on a scale | 56.3 (10.40) | 56.2 (10.28)

16. Other Pre Specified Outcome: Baseline Urge to Cough Questionnaire (UtCQ) 100 mm Visual Analogue Scale
Description: UtCQ is determined through the use of a 100mm visual analogue scale (VAS) (ranging between 0 for "no urge to cough" and 100 for "severe urge to cough").
Time Frame: Baseline (Day 0) of each study period
Population: Analysis population consisted of all participants for Periods 1 and 2 who were randomized, were compliant with the study procedure and had available data at baseline for UtCQ.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Gefapixant 600 mg | Placebo
Number analyzed (Participants) | 24 | 20
Score on a scale | 63.1 (23.10) | 62.5 (19.99)

ADVERSE EVENTS:
Time Frame: Up to 59 days
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a study drug that does not necessarily have a causal relationship and is related or not related to the administration of the study drug or treatment.
Arm/Group | Gefapixant 600 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 24/24 | 5/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant 600 mg (N=24) | Placebo (N=22)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Anosmia (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 21 (21) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (2)
Hypogeusia (Nervous system disorders) | 13 (13) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical trial are the property of Sponsor and are confidential. Authorship on any publication or presentation of the results from this study will be govern by the executed Clinical Trial Agreement as well as being consistent with the Uniform Requirements of the International Committee of Medical Journal Editors.